CLINICAL TRIAL: NCT05531747
Title: Replicative Stress in Hair Follicle Stem Cells and Pathogeny of Hidradenitis Suppurativa
Acronym: Fol-Hydra
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP211351
Record Dates: First submitted 2022-06-14; First posted 2022-09-08 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Hidradenitis Suppurativa
Keywords: cytokine; inflammation; replicative stress; Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Masking Description: Biological assays will be performed by technician blinded from patients clinical status
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physiopathologic exploration (Experimental): A non randomised study with one arm, addind experimental acts to standard of care (skin biopsy and biological sample ) in order to explore Hidradenitis Suppurativa physiopathology
  Interventions: Other: Skin biopsy; Other: Blood sample

INTERVENTIONS:
Other: Skin biopsy — A maximum of 2 superficial skin biopsies (epidermis/dermis), allowing 10 hair follicles to be obtained, at the edge of the affected area, in healthy territory (excluding the face and folds but not excluding the pubic region), at initiation visit.
Other: Blood sample — 42mL of blood (6 tubes of 7mL) sampled at initiation visit

SUMMARY:
Hidradenitis Suppurativa is a recurrent chronic inflammatory follicular occlusive disease affecting hair follicles. HS is notoriously difficult and challenging to treat with a high morbidity impact and could be classified as an unmet medical need with no efficient therapeutic options.

Objective:

Investigators previously showed that Outer Root Sheath Cells (ORS) isolated from hair follicle of HS patients (HS-ORS) have a pro-inflammatory phenotype and secrete spontaneously IP-10 and RANTES. To identify the mechanisms involved in the pro-inflammatory phenotype of HS-ORS, investigators performed a transcriptomic analysis in healthy and HS patients. This revealed: (i) an IFN signature, (i) a dysregulation of genes involved in cell proliferation and differentiation, and (iii) an upregulation of DNA damage response and cell cycle G2/M checkpoint pathways in HS-ORS. These findings support the notion that, in HS patients, a perturbation of HF-SC homeostasis leading to an increased proliferation induces a replicative stress and an accumulation of cytoplasmic ssDNA, stimulating IFN synthesis through IFI16-STING pathway. Interestingly, replicative stress in ORS were present in some but not all patients with Hidradenitis Suppurativa. The goal of study is to determine replicative stress in ORS in a large cohort of HS patients.

Method Patients will be enrolled in the Mondor Dermatology department, during routine care. A dermatologist will check all inclusion and exclusion criteria with the technical support of a research technician of the Henri Mondor Clinical Investigation Center. Medical history, clinical data, comorbidities and concomitant therapies will be prospectively recorded in a dedicated case report form. Skin biopsies will be performed in perilesional zone rich in hair follicles. mRNA will be extracted from freshly isolated hair follicle cells and some slides will be prepared and stored at -80°C to perform immunohistochemistry analysis on freshly isolated hair follicle cells. PBMC and serum will be collected.

All these biological samples will allow us to quantify the replicative stress in HS-ORS of each patient, and to quantify several cytokine of interest : IFN de type 1, IL-17, IL-6, TNF-α, IL-10

This study will allow investigators to evaluate the rate of patients with replicative stress in hair follicle stem cells in Hidradenitis Suppurativa. The investigator will also determine whether HF-SC replication stress correlates with clinical characteristics and/or with clinical course and/or comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the consultation of dermatology of Henri Mondor Hospital
* Diagnosis of Hidradenitis Suppurativa
* Age> 18 y.o.
* Affiliation to a social security system

Exclusion Criteria:

* Patient under tutorship or curatorship
* Breastfeeding or pregnant women
* Refusal to sign the consent letter
* Patients benefiting from State Medical Aid

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2029-06-13 (Estimated); Study Completion 2029-12-13 (Estimated)

PRIMARY OUTCOMES:
Replicative stress in hair follicle stem cells in Hidradenitis Suppurativa | The primary outcome will be evaluated at baseline
  Evaluation of the rate of patients with replicative stress in hair follicle stem cells in Hidradenitis Suppurativa

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU Henri Mondor, Créteil, Val-de-marne, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION